CLINICAL TRIAL: NCT06260228
Title: HOme-Based Self-management and COgnitive Training CHanges Lives (HOBSCOTCH)-Parkinson's Disease (HOBSCOTCH-Parkinson's)
Acronym: HOBSCOTCH-PD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Elaine T. Kiriakopoulos, Assistant Professor of Neurology, Geisel School of Medicine at Dartmouth Director, HOBSCOTCH Institute for Cognitive Health & Well-Being Dartmouth Hitchcock Epilepsy Center, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY02002270
Record Dates: First submitted 2024-01-29; First posted 2024-02-15 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Parkinson Disease; Cognitive Dysfunction; Memory Disorders
Keywords: Parkinson Disease; Memory; Cognitive Training; Self-Management
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction; Memory Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD Participant with Cognitive Dysfunction (Other): Participants will receive the HOBSCOTCH-PD intervention consisting of 1:1 sessions delivered once per week including:
  * 1 pre-HOBSCOTCH Session (on webcam or by phone)
  * 1 educational session (on webcam)
  * 6 HOBSCOTCH intervention sessions (webcam or phone)
  * 1 wrap-up session (webcam or phone)
  Interventions: Behavioral: HOme-Based Self-management and COgnitive Training CHanges lives (HOBSCOTCH)

INTERVENTIONS:
Behavioral: HOme-Based Self-management and COgnitive Training CHanges lives (HOBSCOTCH) — HOBSCOTCH is a home-based self-management program to treat cognitive symptoms and improve quality of life, while minimizing the barriers of access to care. The program is based on Problem Solving Therapy (PST) and teaches problem solving strategies and compensatory mechanisms to help manage cognitive dysfunction and enhance quality of life. HOBSCOTCH-PD is an adaptation of the HOBSCOTCH program for people with PD and incorporates education about Parkinson Disease and cognition into the education module.
  Other Names: HOBSCOTCH-PD

SUMMARY:
The goal of this pilot study is to assess the feasibility of adapting and delivering the existing home-based epilepsy self-management intervention, HOBSCOTCH, for people with Parkinson's Disease (PD)

The main questions it aims to answer are:

1. Can the current HOBSCOTCH program be adapted for people with PD?
2. Will people with PD experience improved quality of life similar to that found in people with epilepsy after participating in the HOBSCOTCH program?

Participants will be asked to:

* attend nine, one-hour virtual (online and/or by telephone) HOBSCOTCH-PD sessions with a one-on-one certified HOBSCOTCH-PD coach
* complete a brief clinical questionnaire about their diagnosis of PD
* complete two questionnaires before and after the HOBSCOTCH-PD sessions about their quality of life and about memory and thinking processes
* keep a short daily diary about their PD symptoms and use of the self-management strategies taught in the HOBSCOTCH-PD program
* complete a brief Satisfaction Survey after the entire HOBSCOTCH-PD program

ELIGIBILITY:
Inclusion Criteria:

* Age 30 - 75 years
* Diagnosis of Parkinson's Disease per participant's provider
* Literate, English-speaking with grade 12 or equivalent in education
* Self-reported cognitive/memory difficulties
* Telephone and internet access

Exclusion Criteria:

* Cognitive dysfunction that precludes participation in giving informed consent
* Significant visual impairment precluding reading or writing
* No reliable telephone or internet access

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2025-09-26 (Actual); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life as measured by comparing PDQ-39 (Parkinson's Disease Questionnaire) scores pre- and post-HOBSCOTCH-PD intervention. | Baseline (pre-HOBSCOTCH-PD) and post-HOBSCOTCH-PD, approximately 9 weeks later.
  The Parkinson's Disease Questionnaire (PDQ-39) is a 39-item validated, patient reported measure of quality of life. The questionnaire assesses how often people with PD experience difficulties across 8 dimensions of daily living including relationships, social situations and communication as well as the impact of Parkinson's on specific dimensions of functioning and wellbeing. The dimension scores are coded on a scale of 0 (perfect health as assessed by the measure) to 100 (worst health as assessed by the measure).
Change in subjective cognition as measured by comparing Neuro-QOL Item Bank v2.0 Cognitive Function scores pre- and post-HOBSCOTCH-PD intervention. | Baseline (pre-HOBSCOTCH-PD) and post-HOBSCOTCH-PD, approximately 9 weeks later.
  The Cognitive Function sub-scale of the Neuro-QOL is a brief validated tool developed by the NIH for use in patients with neurological disease. Scores range from 8 to 40, with a higher score indicating better reported cognitive functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine T Kiriakopoulos, MD, MPH, MSc, Principal Investigator — Dartmouth-Hitchcock, Dartmouth College
Locations (1):
- Dartmouth-Hitchcock, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No